CLINICAL TRIAL: NCT04577170
Title: Association of the Pulsatility Index and Vasomotor Reactivity With White Matter Lesions in Brain MRI of Fabry Disease Patients
Brief Title: Pulsatility Index, Vasomotor Reactivity and Leukoencephalopathy in Fabry Patients
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Georgios Tsivgoulis, Professor, National and Kapodistrian University of Athens
Other Study IDs: FD29092020
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Fabry Disease
Keywords: pulsatility index; vasomotor reactivity; leukoencephalopathy; transcranial ultrasound
MeSH Terms: conditions — Fabry Disease; Leukoencephalopathies | interventions — Ultrasonography, Doppler, Transcranial; Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fabry disease
  Interventions: Diagnostic Test: Transcranial Doppler (TCD) and Transcranial Color-Coded Duplex (TCCD) ultrasonography
- Healthy: age and sex matched
  Interventions: Diagnostic Test: Transcranial Doppler (TCD) and Transcranial Color-Coded Duplex (TCCD) ultrasonography

INTERVENTIONS:
Diagnostic Test: Transcranial Doppler (TCD) and Transcranial Color-Coded Duplex (TCCD) ultrasonography — Transcranial Doppler (TCD) and Transcranial Color-Coded Duplex (TCCD) ultrasonography will be performed in consecutive FD patients. All TCD and TCCD studies will be performed by stroke neurologists experienced in vascular sonography.

SUMMARY:
We hypothesize that Fabry disease - FD is associated with elevated vascular resistance induced by cerebral small-vessel disease, indicating increased distal resistance to blood flow. The findings of this study may be used as a precursor for neuroimaging manifestations related to stroke in FD patients.

ELIGIBILITY:
Inclusion Criteria:

Fabry disease diagnosis, genetically confirmed Age> 16 years

Exclusion Criteria:

Insufficient temporal bone window MRI contra-indication Inability to cooperate for breath-holding test Detection of atrial fibrillation Refuse to sing informed consent

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with genetically confirmed FD and healthy individuals will be prospectively enrolled as part of routine clinical examination.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of elevated pulsatility index of FD patients | 2 years
  to assess the prevalence of elevated pulsatility index in FD patients at a single time point.
Prevalence of elevated vasomotor reactivity in FD patients. | 2 years
  to assess the prevalence of elevated vasomotor reactivity in FD patients at a single time point.

SECONDARY OUTCOMES:
Association of pulsalitily index with leukoencephalopathy in FD patients. | 2 years
  To associate the pulsality index measured by TCD and TCCD with the presence of white matter lesions in brain MRI of FD patients.
Association of vasomotor reactivity with leukoencephalopathy in FD patients. | 2 years
  To associate the vasomotor reactivity measured by TCD and TCCD with the presence of white matter lesions in brain MRI of FD patients.
Τo compare the pulsatility index measured in FD patients against corresponding prospectively collected data from healthy individuals, stratified by age and sex. | 2 years
  For the secondary outcome, age and sex-matched healthy controls will be consecutively enrolled. After clinical evaluation, healthy controls will present no FD-associated manifestations, hence they will be FD negative. In addition, brain MRI will be performed and subjects with white matter disease and leukoencephalopathy will be excluded. Included controls will be leukoencephalopathy negative. TCD and TCCD evaluation will be performed in healthy controls, in order to measure pulsatility index and compare the results against FD patients.
Τo compare vasomotor reactivity measured in FD patients against corresponding prospectively collected data from healthy individuals, stratified by age and sex. | 2 years
  For the secondary outcome, age and sex-matched healthy controls will be consecutively enrolled. After clinical evaluation, healthy controls will present no FD-associated manifestations, hence they will be FD negative. In addition, brain MRI will be performed and subjects with white matter disease and leukoencephalopathy will be excluded. Included controls will be leukoencephalopathy negative. TCD and TCCD evaluation will be performed in healthy controls, in order to measure vasomotor reactivity and compare the results against FD patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Department of Neurology, "Attikon" University Hospital, School of Medicine, National and Kapodistrian University of Athens, Athens, Greece, Athens, Greece